CLINICAL TRIAL: NCT04432259
Title: Oral Dexamethasone as an Intervention for Postoperative Pain and Nausea Management in Total Knee Arthroplasty
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Jonathan H. Shaw, Orthopaedic Surgeon, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13565
Record Dates: First submitted 2020-06-12; First posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Arthritis Knee; Postoperative Nausea; Postoperative Pain
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Pain, Postoperative | interventions — Dexamethasone

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two groups, treatment or no treatment. Randomizations will be balanced at random accrual points.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm B: Oral Dexamethasone (Experimental): Participants will be randomly assigned to receive 4 mg Oral Dexamethasone taken twice daily for 4 days
  Interventions: Drug: Dexamethasone
- Arm A: Placebo (Placebo Comparator): Participants will be randomly assigned to receive 4 mg placebo taken twice daily for 4 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexamethasone — 4 mg bid for 4 days
  Arms: Arm B: Oral Dexamethasone
Drug: Placebo — oral placebo
  Arms: Arm A: Placebo

SUMMARY:
This study aims to determine if oral dexamethasone provides clinically significant improvement in postoperative outcomes, specifically nausea and pain scores.

DETAILED DESCRIPTION:
Protocols in perioperative pain management during total joint arthroplasty (TJA) have contributed to early discharge after surgery. As practices move to favor ambulatory surgery in total joint arthroplasty changes must be made to postoperative pain and nausea management. Spinal anesthesia has been essential in managing associated ambulatory TJA, however, nausea and vomiting are known detrimental side effects. The use of systemic steroids has also been shown in the literature to reduce pain scores, length of stay, the need for antiemetics, and increase the distance of ambulation without increasing the rate of surgical site infection or prosthetic joint infection. As more same-day total joint replacement is incorporated into practice, an oral alternative may prove beneficial.

ELIGIBILITY:
Inclusion Criteria:

* adult patients age 18 and older who will be undergoing joint replacement

Exclusion Criteria:

* Patients with uncontrolled diabetes ( HbA1C, >7.5%), impaired hepatic function (Child class, >B), impaired renal failure (Glomerular filtration rate <60 mL/min/1.73 m2), chronic narcotic use, alcohol and/or opioid dependence, patients with a known adverse reaction to corticosteroids, and patients unable to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-07 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain | 3 weeks following surgery
  Postoperative pain will be collected via visual analog scores
Postoperative Nausea | 3 weeks following surgery
  Postoperative Nausea will be collected via visual analog scores
Opioid Consumption | 6 months
  Opioid consumption will be recorded by participant in assigned journal, morphine equivalence will be recorded
Antiemetic Consumption | 6 months
Episodes of Nausea | 3 weeks

SECONDARY OUTCOMES:
Postoperative complications | 6 months
  Incidence of surgical site infection, acute prosthetic joint infection
Patient-reported outcome scores (PROMS) | 6 months
Knee Injury and Osteoarthritis Outcome Score (KOOS) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jason Davis, M.D., Principal Investigator — Henry Ford Health System